CLINICAL TRIAL: NCT04913077
Title: Prospective One-armed Observational Study of Full-thickness Resection of Small Hypoechoic Submucosal Gastric Tumors (≤2 cm)
Brief Title: Submucosal Tumor Removal by Endoscopic Excision Therapy
Acronym: STREET
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: interim analysis
Sponsor: Universitätsklinikum Hamburg-Eppendorf (Other)
Collaborators: Ovesco Endoscopy AG (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: PV7129
Record Dates: First submitted 2021-01-23; First posted 2021-06-04 (Actual); Last update posted 2024-03-19 (Actual); Status verified 2024-03

CONDITIONS: Submucosal Tumor of Stomach
Keywords: Submucosal Tumor of Stomach; GIST; FTRD
MeSH Terms: interventions — Endoscopic Mucosal Resection

STUDY DESIGN:
Intervention Model Description: Submucosal gastric Tumors up to 2 centimeters of size
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Removal of submucosal gastric tumor preferably by Full Thickness Resection Device (FTRD) (Other): FTRD (Ovesco company) in tumors up to 10 mm and predominantly intraluminal growth directly by sucking into the cap, at 10-20 mm and/or intramural/extramural growth by prior circumcision and lateral preparation, so that the lesions can be better pulled into the cap. The procedure depends on the endosonographic extent of the findings. The lesions are pulled into the cap with grippers and other instruments and, if necessary, with a snare and then resected with FTRD
  Interventions: Other: removal of submucosal gastric tumor preferably by Full Thickness Resection Device (FTRD)

INTERVENTIONS:
Other: removal of submucosal gastric tumor preferably by Full Thickness Resection Device (FTRD) — FTRD (Ovesco company) in tumors up to 10 mm and predominantly intraluminal growth directly by sucking into the cap, at 10-20 mm and/or intramural/extramural growth by prior circumcision and lateral preparation, so that the lesions can be better pulled into the cap. The procedure depends on the endosonographic extent of the findings. The lesions are pulled into the cap with grippers and other instruments and, if necessary, with a snare and then resected with FTRD
  Other Names: Endoscopic submucosal dissection (ESD)

SUMMARY:
Smaller submucosal tumors (SMT) in the stomach are usually seen as an incidental finding during a gastroscopy, although current diagnostics usually do not clearly indicate what type of tumor it is. In summary, there is no good evidence for dealing with SMT. In this study, an endoscopic full-thickness resection, primarily with the FTRD device, is to be offered to all patients with gastric SMT without a confirmed histology seen in a certain period of time . Patients who do not want to take advantage of this are included in a systematic follow-up program.

The investigators hope to learn about the rate of so-called GIST tumors and other histologies, as well as the rate of change in the follow-up group.

Also, study contents will be accuracy of endosonographic imaging and puncture in comparison with resection histology, technical feasibility and histological completeness of the FTRD- based endoscopic (full-wall) resection option, complications of such a resection (secondary bleeding and dehiscences), and patient preferences with standardized information.

DETAILED DESCRIPTION:
Smaller submucous tumors in the stomach are usually seen as a random finding in gastroscopies and present a diagnostic dilemma to the doctor and patient:

type specification is usually unclear whether it is an absolutely benign (without degeneration potential) or a malignant or prone tumor (usually gastrointestinal stromal tumor, GIST). However, this is crucial for further management.

In endosonographic imaging there are only approximate values in the differential diagnosis between GIST and non-GIST, the endoscopic biopsy is too superficial, and the hit rate of endosonographic pin puncture is limited, and in most studies is less than 70% Therefore, one can only make assumptions and create a risk profile from imaging and tumor size (limit size 3 cm, partly also 2 cm). Both follow-up recommendations (rather no GIST) and laparoscopic surgical removal (proven or probable/possible GIST) are not rarely without clear preference, especially for smaller tumors.

For these indications, a simple endoscopic removal option comparable to the polypectomy in the colon (where no histological type diagnosis is made before) does not exist.

Previous studies are usually subject to bias in several directions:

1. The frequency of GIST tumors among submucous tumors/lesions (SMT) in the stomach is unclear. Gastroenterological series always contain smaller GIST tumors, but are reported almost exclusively from clinics. The rate of these tumors in the overall collective of patients seen in the field of (mostly established) gastroenterologists is thus completely unclear. Surgical or oncological series have usually included more aggressive tumors consisting mainly or exclusively of GIST tumors, therefore do not allow epidemiological conclusions.
2. If no surgery is performed (and thus a definitive histology is forced), only information from follow-up examinations remains. Previous follow-up studies show the dilemma of insufficient differential diagnosis of lesions by endosonography and (endosonographic or other) biopsy, which usually have insufficient accuracy. In addition, the follow-up time in the studies hardly extends beyond 2 years. The "gastroenterological gut instinct" that these small lesions are not dangerous may be true, but is not proven.

ELIGIBILITY:
Inclusion Criteria:

* Patients with endoscopically diagnosed and endosonographically confirmed submucosal tumors of 0.5 to 2 cm in the stomach without definitive histology / cytology
* Initial diagnosis less than 2 years ago
* No contraindication to endoscopic resection
* Patient's informed consent

Exclusion Criteria:

* Tumor size > 2 cm
* Tumors with proven / suspected malignancy for which oncologically no endoscopic resection should be performed, i.e. for which oncological or surgical therapy is planned
* SMT known > 2 Years
* Patients with severe general illnesses (limited operability) or malignancies
* Clotting disorders
* Pregnancy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2020-03-10 (Actual); Primary Completion 2024-11 (Estimated); Study Completion 2025-02 (Estimated)

PRIMARY OUTCOMES:
Rate of GIST tumors | through study completion, approximately 2 years
  Rate of GIST tumors in a preferably unselected patient cohort of small submucous gastric tumors in which histology is not known

SECONDARY OUTCOMES:
Technical success | through study completion, approximately 2 years
  Technical success rate (R0/R1 resection) of the chosen resection technique
Complication rate | through study completion, approximately 2 years
  Complication rate of the chosen resection technique
influencing factors on the GIST rate: tumor size | through study completion, approximately 2 years
  Influence of tumor size on the GIST rate
Influencing factors on the GIST rate: position of tumor | through study completion, approximately 2 years
  Influence of tumor position in the stomach
Influencing factors on the GIST rate: endoscopic ultrasound image | through study completion, approximately 2 years
  endoscopic ultrasound image with pattern and position in the wall
Influencing factors on the GIST rate: patient's age | through study completion, approximately 2 years
  Age of patients
Influencing factors on the GIST rate: patient's gender | through study completion, approximately 2 years
  gender of patients
Influencing factors on the GIST rate: anamnesis | through study completion, approximately 2 years
  anamnesis including initial diagnosis
Patient's preferred approach | through study completion, approximately 2 years
  Patient preferences for removal (consent rate for the study) versus follow-up
data for cost-benefit calculation | through study completion, approximately 2 years
  Establishment of a date base for a cost-benefit calculation comparing follow-up vs. removal

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Rösch, Prof. Dr., Principal Investigator — Universitätsklinikum Hamburg-Eppendorf
Locations (3):
- Germany (3):
  - University Hospital Freiburg, Freiburg im Breisgau
  - University Hospital Hamburg Eppendorf, Hamburg
  - University Hospital Marburg, Marburg

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cai MY, Martin Carreras-Presas F, Zhou PH. Endoscopic full-thickness resection for gastrointestinal submucosal tumors. Dig Endosc. 2018 Apr;30 Suppl 1:17-24. doi: 10.1111/den.13003. PMID 29658639
- [Background] Akahoshi K, Oya M, Koga T, Shiratsuchi Y. Current clinical management of gastrointestinal stromal tumor. World J Gastroenterol. 2018 Jul 14;24(26):2806-2817. doi: 10.3748/wjg.v24.i26.2806. PMID 30018476
- [Background] Cazacu IM, Luzuriaga Chavez AA, Nogueras Gonzalez GM, Saftoiu A, Bhutani MS. Malignant Transformation of Ectopic Pancreas. Dig Dis Sci. 2019 Mar;64(3):655-668. doi: 10.1007/s10620-018-5366-z. Epub 2018 Nov 10. PMID 30415408
- [Background] Standards of Practice Committee; Faulx AL, Kothari S, Acosta RD, Agrawal D, Bruining DH, Chandrasekhara V, Eloubeidi MA, Fanelli RD, Gurudu SR, Khashab MA, Lightdale JR, Muthusamy VR, Shaukat A, Qumseya BJ, Wang A, Wani SB, Yang J, DeWitt JM. The role of endoscopy in subepithelial lesions of the GI tract. Gastrointest Endosc. 2017 Jun;85(6):1117-1132. doi: 10.1016/j.gie.2017.02.022. Epub 2017 Apr 3. No abstract available. PMID 28385194
- [Background] Kida M, Kawaguchi Y, Miyata E, Hasegawa R, Kaneko T, Yamauchi H, Koizumi S, Okuwaki K, Miyazawa S, Iwai T, Kikuchi H, Watanabe M, Imaizumi H, Koizumi W. Endoscopic ultrasonography diagnosis of subepithelial lesions. Dig Endosc. 2017 May;29(4):431-443. doi: 10.1111/den.12854. Epub 2017 Apr 6. PMID 28258621
- [Background] Kim SY, Kim KO. Management of gastric subepithelial tumors: The role of endoscopy. World J Gastrointest Endosc. 2016 Jun 10;8(11):418-24. doi: 10.4253/wjge.v8.i11.418. PMID 27298713
- [Background] Kim SY, Kim KO. Endoscopic Treatment of Subepithelial Tumors. Clin Endosc. 2018 Jan;51(1):19-27. doi: 10.5946/ce.2018.020. Epub 2018 Jan 31. PMID 29397653
- [Background] Lim TW, Choi CW, Kang DH, Kim HW, Park SB, Kim SJ. Endoscopic ultrasound without tissue acquisition has poor accuracy for diagnosing gastric subepithelial tumors. Medicine (Baltimore). 2016 Nov;95(44):e5246. doi: 10.1097/MD.0000000000005246. PMID 27858880
- [Background] Marcella C, Shi RH, Sarwar S. Clinical Overview of GIST and Its Latest Management by Endoscopic Resection in Upper GI: A Literature Review. Gastroenterol Res Pract. 2018 Oct 31;2018:6864256. doi: 10.1155/2018/6864256. eCollection 2018. PMID 30515204
- [Background] Moon JS. Role of Endoscopic Ultrasonography in Guiding Treatment Plans for Upper Gastrointestinal Subepithelial Tumors. Clin Endosc. 2016 May;49(3):220-5. doi: 10.5946/ce.2016.047. Epub 2016 May 20. PMID 27209643
- [Background] Bruno M, Carucci P, Repici A, Pellicano R, Mezzabotta L, Goss M, Magnolia MR, Saracco GM, Rizzetto M, De Angelis C. The natural history of gastrointestinal subepithelial tumors arising from muscularis propria: an endoscopic ultrasound survey. J Clin Gastroenterol. 2009 Oct;43(9):821-5. doi: 10.1097/MCG.0b013e31818f50b8. PMID 19349904
- [Background] Kim MY, Jung HY, Choi KD, Song HJ, Lee JH, Kim DH, Choi KS, Lee GH, Kim JH. Natural history of asymptomatic small gastric subepithelial tumors. J Clin Gastroenterol. 2011 Apr;45(4):330-6. doi: 10.1097/MCG.0b013e318206474e. PMID 21278578
- [Background] Kushnir VM, Keswani RN, Hollander TG, Kohlmeier C, Mullady DK, Azar RR, Murad FM, Komanduri S, Edmundowicz SA, Early DS. Compliance with surveillance recommendations for foregut subepithelial tumors is poor: results of a prospective multicenter study. Gastrointest Endosc. 2015;81(6):1378-84. doi: 10.1016/j.gie.2014.11.013. Epub 2015 Feb 7. PMID 25660977